CLINICAL TRIAL: NCT07094256
Title: Evaluation of Novel Torque Device During Electrophysiology Study Procedure
Brief Title: Torque Device Evaluation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PEDS-2024-33423
Record Dates: First submitted 2025-07-22; First posted 2025-07-30 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Electrophysiology Study; Ablation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Torque Device (Experimental): After the completion of the electrophysiology study and/or ablation procedure, the catheters remain in the intra-cardiac locations. While in place, measurements will be obtained from each catheter. Once the baseline measurements have been obtained, the Peritorq device will be placed onto each relevant catheter. Once secured, all measurements will be repeated with each catheter at the identical location. After measurements have been obtained, the operator will perform minor catheter movements to note subjective maneuverability and stability of the catheter with the torque device in place
  Interventions: Device: Peritorq

INTERVENTIONS:
Device: Peritorq — Novel torque device specifically designed for electrophysiology and ablation catheters

SUMMARY:
This study will evaluate the safety and efficacy of a novel catheter torque device after the completion of a clinically-indicated electrophysiology study and/or ablation procedure in a pediatric patient. All electrophysiology studies and/or ablation procedures will be performed at the discretion of their primary cardiologist and will not be affected by this study protocol. The study protocol will commence once the attending electrophysiologist has completed all necessary intervention and testing and no further evaluation is required.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient (≤21 years of age)
* Undergoing clinically-indicated electrophysiology study and/or ablation procedure

Exclusion Criteria:

* Adult patient (>21 years)

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Difference in Impedance | 15 minutes
  Obtained from catheter at baseline and after Peritorq device placed
Difference in Sensing of Chamber Amplitude (mV) | 15 minutes
  Obtained from catheter at baseline and after Peritorq device placed
Difference in Capture Threshold of Atrium and Ventricle (mA) | 15 minutes
  Obtained from catheter at baseline and after Peritorq device placed

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No